CLINICAL TRIAL: NCT06858124
Title: Comparison of Mulligan and Maitland Mobilization Techniques Combined With Home-Based Exercise for Non-Specific Neck Pain: A Randomized Controlled Trial
Brief Title: Mulligan vs Maitland With Home-Based Exercise for Non-Specific Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Hellenic University (Other)
Responsible Party: Principal Investigator, Dimitrios Lytras, Assistant Professor, International Hellenic University
Allocation: Not Applicable | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC-5/2025
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Neck Pain
Keywords: Non-Specific Neck Pain; Mulligan; Maitland
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: 43 participants with non-specific neck pain pain will be randomly assigned to three groups of 14, 14 and 15 participants each. The allocation of the sample to the groups will be performed using the randomization app Randomiser (Rob Sammons, Apple Store) by an independent researcher. In the first group, a mulligan mobilization protocol will be applied and the practitioners will follow a daily therapeutic exercise program at home, in the second group, a maitland mobilization protocol will be applied and the practitioners will follow a daily therapeutic exercise program at home, while the third group will follow only a daily therapeutic exercise program at home. Participants of the two intervention groups will follow a total of four treatments over a period of two weeks. The therapeutic home-based exercise program will be performed daily over the same period of two weeks.
Who Masked: Care Provider
Masking Description: A masked assessor will conduct the measurements
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mulligan+TE (Experimental): Participants allocated to this group will receive four sessions of Mulligan mobilizations and will perform a home-based therapeutic exercise program for two weeks.
  Interventions: Other: Mulligan+TE
- Maitland +TE (Experimental): Participants allocated to this group will receive four sessions of Maitland mobilizations and will perform a home-based therapeutic exercise program for two weeks.
  Interventions: Other: Maitland+TE
- Active Comparator: "TE group". (Active Comparator): Participants in this group will only perform the same 4 home-based therapeutic exercises as the first group.

INTERVENTIONS:
Other: Mulligan+TE — Mulligan Mobilizations plus Home Therapeutic Exercise
  The protocol will last 25 minutes (Mulligan protocol: 5 minutes and Home Therapeutic Exercise protocol: 20 minutes) and will include the application of the following mulligan techniques and home exercises:
  * Mulligan sustained natural apophyseal glide SNAG mobilizations with overpressure with the patients in seated position.
  * 4 home-based therapeutic exercises: isometric exercises for cervical regions, head retractions, thoracic spine rotation mobility exercise and diagonal cervical mobility exercise pattern.
  Arms: Mulligan+TE
Other: Maitland+TE — The participants of this group will perform the same 4 home-based therapeutic exercises as the first group. In addition, they will receive a 5-minute maitland mobilization protocol.
  Maitland mobilizations will include posterioranterior glides with oscillations with the patients in prone position.
  Arms: Maitland +TE
Other: Control — Participants in this group will only perform the same 4 home-based therapeutic exercises as the first group.

SUMMARY:
Non-specific neck pain (NSNP) is a prevalent musculoskeletal condition with multiple contributing factors. The aim of this clinical study is to investigate the short-term effects of Mulligan in comparison to Maitland mobilization techniques in conjunction with a home-based therapeutic exercise program. 43 adults with non-specific neck pain will be randomly divided into three groups of 14,14 and 15 participants each. In the participants of the first group, a therapeutic protocol of Mulligan mobilizations in the cervical region will be applied and a protocol of exercises will be performed. To the participants of the second group, a therapeutic protocol od Maitland mobilizations in the cervical region will be applied and the same exercise program with the first group will be performed. The third group participants will perform only the same exercise protocol as the other groups. The first two groups will receive four mobilization treatments over two weeks. All three groups will perform the home-based exercise protocol daily for two weeks. Pain in the last 24 hours with the Numeric Pain Rating Scale (NPRS), Pressure Pain Threshold (PPT) in the cervical region with an algometer, functional ability with the Neck Disability Index (NDI), Range of Motion (ROM) with a digital goniometer, pain catastrophizing with the Pain Catastrophizing Scale (PCS) and kinesiophobia with the Tampa Scale of Kinesiophobia (TSK) will be evaluated before and after the intervention. For the statistical analysis of the results, a two-way repeated measures analysis of variance (ANOVA) will be applied using SPSS program, while the statistical significance index will be set at p < .05.

DETAILED DESCRIPTION:
Background: Non-specific neck pain (NSNP) is a prevalent musculoskeletal condition with multiple contributing factors. Various manual therapy approaches, such as Mulligan and Maitland mobilizations, are commonly applied to alleviate pain and enhance function.

Aim: The purpose of this clinical study is to investigate the short-term effects of Mulligan in comparison to Maitland mobilization techniques in conjunction with a home-based therapeutic exercise (TE) program.

Method: 43 participants with non-specific neck pain will be randomly assigned to three groups of 14, 14 and 15 participants each. In the participants of the first group, a therapeutic protocol of mulligan mobilizations will be applied to the cervical region. In addition, the participants will perform a home-based therapeutic exercise program. To the participants of the second group, a therapeutic protocol of maitland mobilizations will be applied to the cervical region and they will perform the same home-based exercise protocol with the first group. The third group participants will perform only the same home-based exercise protocol with the other groups. The first two groups will receive four mobilization treatments over two weeks. All three groups will perform the home-based exercise protocol daily for two weeks. Pain in the last 24 hours with the Numeric Pain Rating Scale (NPRS), Pressure Pain Threshold (PPT) in the cervical region with an algometer, functional ability with the Neck Disability Index (NDI), Range of Motion (ROM) with a digital goniometer, pain catastrophizing with the Pain Catastrophizing Scale (PCS) and kinesiophobia with the Tampa Scale of Kinesiophobia (TSK) will be evaluated before and after the intervention. For the statistical analysis of the results, a two-way repeated measures analysis of variance (ANOVA) will be applied using SPSS program, while the statistical significance index will be set at p < .05. Expected results: The protocol proposed in this clinical study combines the benefits of applying manual therapy mobilizations with the beneficial effects of therapeutic exercise. Previous research shows Mulligan mobilizations may be slightly more beneficial in improving patients' symptoms with non-specific neck pain. For this reason, we expect that the combination of Mulligan mobilizations and home-based therapeutic exercise will be more effective than the combination of Maitland mobilizations and home-based therapeutic exercise only in improving the clinical symptoms of young adults with non-specific neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Acute-subacute-chronic neck pain
* Women - Men
* Age range between 18 and 30 years
* NPRS score >2
* Written consent to participate in the study

Exclusion Criteria:

* • Previous cervical/thoracic surgery

  * Recent whiplash (≤6 months)
  * Upper cervical pathology
  * Osteoporosis
  * Pregnancy
  * Cancer
  * Systemic diseases or spinal disorders
  * Neurological symptoms
  * Severe medical conditions, positive red flags (Spurling test, Hoffmann's sign, Babinski reflex, clonus)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2025-02-27 (Actual); Primary Completion 2025-04-05 (Actual); Study Completion 2025-04-05 (Actual)

PRIMARY OUTCOMES:
Changes in neck pain intensity with Numeric Pain Rating Scale (NPRS) | pre-treatment, week: 2
  This tool is an 11-point scale from 0 ("no pain") to 10 ("worst imaginable pain"). Consequently, a higher value indicates more intense pain. The participant selects a number that best represents their pain intensity. The NPRS is a well-validated tool commonly used to measure pain intensity in clinical practice and research.
Changes in Pressure Pain Threshold (PPT) with pressure algometry | pre-treatment, week: 2
  Pressure pain threshold (PPT) is defined as the minimal amount of pressure that produces pain. PPT will be assessed by a digital algometer and will be evaluated bilaterally in the upper trapezius muscle, between C7 and the acromion. The rubber tip of the algometer will be placed vertically on the site and the examiner will apply gradually increasing pressure in a rate of 1Kg/s.
Changes in cervical range of motion with digital goniometry | pre-treatment, week: 2
  The cervical ROM of cervical flexion, extension, side bends and rotations will be assessed using a digital goniometer with the patient in the seated position. Each movement will be carried out once within the maximum pain-free range and will be documented by an independent physiotherapist
Changes in functional ability with Neck Disability Index (NDI) | pre-treatment, week: 2]
  The Neck Disability Index (NDI), validated for the Greek population, will be used to assess disability. It comprises 10 sections that evaluate pain intensity, functional restrictions, and daily activities, with a total score ranging from 0 (no disability) to 50 (severe disability).
Changes in pain catastrophizing with Pain Catastrophizing Scale (PCS | pre-treatment, week: 2]
  The Pain Catastrophizing Scale (PCS) will be used to assess pain catastrophizing. It is a 13-item questionnaire designed to assess catastrophic thinking related to pain. Scores range from 0 to 52, with higher scores reflecting greater levels of catastrophizing across the subscales of rumination, magnification, and helplessness. The Greek version demonstrates high reliability (ICC = 0.85, Cronbach's α = 0.80).
Changes in kinesiophobia with Tampa Scale of Kinesiophobia (TSK) | pre-treatment, week: 2
  Kinesiophobia will be evaluated using the Tampa Scale of Kinesiophobia (TSK), a 17-item questionnaire that assesses fear of movement and anxiety related to injury. Scores range from 17 to 68, with ≤37 indicating low kinesiophobia and >37 representing high kinesiophobia. The Greek version has demonstrated good reliability (Cronbach's α = 0.74, ICC = 0.78).

CONTACTS AND LOCATIONS:
Locations (1):
- International Hellenic University, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No